CLINICAL TRIAL: NCT00154635
Title: A Double-Blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of DCB-AD1 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety Study of DCB-AD1 in Patients With Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Development Center for Biotechnology, Taiwan (Other Government); Taipei Veterans General Hospital, Taiwan (Other Government); Program Office, National Science & Technology, Biotechnology & Pharmaceuticals (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 931006; NTUH IRB 931006; VGH IRB 93-11-06; DCB-AD1-01-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Dementia, Alzheimer Type
Keywords: Alzheimer's disease; Fo-ti; Chinese herbs
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: DCB-AD1

SUMMARY:
A Double-blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of DCB-AD1 in Patients with Mild to Moderate Alzheimer's Disease. Because of the limitation of the sample size we could expect but a positive trend of the efficacy unless the effect size of DCB-AD1 is larger than 0.63. This information will provide us clue if further clinical investigation such as a phase III study should be carried out in an even larger scale. We also should be able to obtain valuable experience on the adverse effect of prolonged (24-week) use of Fo-ti.

DETAILED DESCRIPTION:
The growing number of patients with dementia has become a great concern of many aging societies. Up to this moment no treatment can stop Alzheimer's dementia (AD), thus, developing new treatments are still mandatory. In this study we will investigate a new drug DCB-AD1, an herbal medicine derived from root of Fo-ti. Historically the Chinese used the Fo-ti root for its rejuvenating properties to treat premature aging, weakness and so on. In DCB (Development Center of Biotechnology)'s preliminary studies using human neuroblastoma cell, SK-N-SH, Fo-ti water extracts exhibited high potential in preventing A-beta and hydrogen peroxide-induced cell death. From two different AD animal models, DCB have observed neuroprotection effects of Fo-ti using water maze and hole-board exploration tests, Though the pharmacological effect of Fo-ti has yet been clarified, its protective effect may result from radical scavenging activities, anti-inflammatory effect or anti-peroxidation. We intend to investigate DCB-AD1 on its cognitive and neurophysiological effects on Alzheimer disease through a randomized, double-blind, placebo-controlled therapeutic trial for 24 weeks. We will complete 80 eligible cases for analysis in this clinical trial with 40 in each investigation site. The estimated drop-out rate is around 25~30 %. Patients are eligible if they fulfill criteria for a diagnosis of probable AD of NINCDS-ADRDA. We will include patients with Mini-Mental State Examination scores of 12~24 and Clinical Dementia Rating 1 or 2. Patients will be allowed to take cholinesterase inhibitors, donepezil, rivastigmine, galantamine or memantine if the dose has been unchanged for the last 3 months before the study entry and remains stable during the 24-week study period.

As for the outcome measures, the primary end point will be the score changes of ADAS-Cog at the end of treatment from the baseline. Secondary end points include CIBIC-PLUS, IADL, Behav-AD, MMSE and CDR.

The statistic analysis will be on both intention-to-treat and completed cases. Because of the limitation of the sample size we would expect but a positive trend of the efficacy unless the effect size of DCB-AD1 is larger than 0.63. This information will provide us clue if further clinical investigation such as a phase III study should be carried out in an even larger scale. We will valuable experience on the adverse effect of prolonged (24-week) use of Fo-ti.

ELIGIBILITY:
Inclusion Criteria:

1. Male or post menopausal female patients aged ≧50 years old;
2. The informed consent must be signed by the patient and co-signed by their proxy or principal caregivers before undergoing any study procedures;
3. Probable Alzheimer's disease based on the National Institute of Neurological and Communicative Disorders and Alzheimer's dementia and related disorder (NINCDS-ADRDA)
4. Patients with Mini-Mental State Examination (MMSE) scores of 12~24
5. Patients with Clinical Dementia Rating (CDR)in mild (CDR = 1) and moderate (CDR = 2) AD
6. Cranial computed tomography (CT) or brain magnetic resonance imaging (MRI) must be within the past 12 months;
7. Patients must be able to complete baseline assessments;
8. An eligible principal caregiver must be able to accompany the patient to all scheduled visits;
9. Patients currently taking ChEIs such as donepezil, rivastigmine, or galantamine are allowed if the dose has been unchanged for the last 3 months before the study entry.

Exclusion Criteria:

1. Patients with history of severe systemic disease such as coronary artery disease, myocardial infarct, progressive heart failure, chronic obstructive pulmonary disease within the past 1 year;
2. Patients with hepatic and renal insufficiency (ALT、AST 3 times above normal range; serum creatinine 2 times above normal range), diabetic patients with poor control of blood sugar (HbA1c>8.5) at study entry;
3. Patients with central nervous system disease other than AD such as cerebral vascular disease, Parkinson's disease, epilepsy, traumatic brain injury, central nervous system infection, and alcoholic encephalopathy;
4. Patients with concurrent psychosis or mood disorder (Hamilton depression scale score > 17);
5. Patients diagnosed cancer and treated within the past two years (except for non-invasive skin cancer);
6. Patients with general medical conditions, which may confound the results of the study, pose additional risk or preclude evaluation and assessments in this study as judged by the investigator;
7. Patients currently treated with any prohibited medications (listed in Concomitant Treatment section) are not able to fulfill the 2 week-washout period;
8. Participation in another study within the last 30 days;
9. Females who are within two years of their menopause unless proved not pregnant (determined by urine test);
10. Dementia caused by other etiology as indicated by clinically significant abnormal Vit B12, folic acid, or thyroid function tests.
11. Patients with neurosyphilis confirmed by CSF STS/TPHA;
12. The neuroimage CT or MRI could not be compatible with the diagnosis of probable AD as stated in the NINCDS criteria;
13. Patients with a Hachinski score (Appendix 5) above 3 are excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-09

PRIMARY OUTCOMES:
ADAS-Cog

SECONDARY OUTCOMES:
CIBIC-PLUS
IADL
Behav-AD
MMSE
CDR

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jang Chiu, MD, PhD, Principal Investigator — NTUH
Locations (2):
- Taiwan (2):
  - NTUH, Taipei, Taipei
  - VGH, Taipei, Taipei